CLINICAL TRIAL: NCT05903339
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Ferritin Nanoparticles Expressing Native-like HIV-1 Envelope Trimers Followed by Boost With mRNA Lipid Nanoparticles Encoding a Native-like HIV-1 Envelope Trimer in Adults Without HIV
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Ferritin Nanoparticles Expressing Native-like HIV-1 Envelope Trimers Followed by Boost With mRNA Lipid Nanoparticles Encoding a Native-like HIV-1 Envelope Trimer in Adults Without HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 307; 38970 (Other: DAIDS DOCUMENT ID)
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — aluminum sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Low dose V3G CH848 Pr-NP1 with 3M-052-AF + Alum (Experimental): 3 doses of V3G CH848 Pr-NP1 (60 mcg) combined with 3M-052-AF (5 mcg) and Alum (500 mcg) at the month 0, 2, and 6 visits, followed by 1 dose of V3G CH848 mRNA-Tr2 (50 mcg) at the month 10 visit
  Interventions: Drug: V3G CH848 Pr-NP1 60mcg; Drug: 3M-052-AF 5mcg; Drug: Alum 500 mcg; Drug: V3G CH848 mRNA-Tr2 50mcg
- Group 2: Low dose V3G CH848 Pr-NP1 with ACU-026-001-1 (Experimental): 3 doses of V3G CH848 Pr-NP1 (60 mcg) combined with ACU-026-001-1 (2.0 mg) at the month 0, 2, and 6 visits, followed by 1 dose of V3G CH848 mRNA-Tr2 (50 mcg) at the month 10 visit
  Interventions: Drug: V3G CH848 Pr-NP1 60mcg; Drug: V3G CH848 mRNA-Tr2 50mcg; Drug: ACU-026-001-1 2.0mg
- Group 3: V3G CH848 Pr-NP1 with 3M-052-AF + Alum (Experimental): 3 doses of V3G CH848 Pr-NP1 (100 mcg) combined with 3M-052-AF (5 mcg) and Alum (500 mcg) at the month 0, 2, and 6 visits, followed by 1 dose of V3G CH848 mRNA-Tr2 (50 mcg) at the month 10 visit
  Interventions: Drug: 3M-052-AF 5mcg; Drug: Alum 500 mcg; Drug: V3G CH848 mRNA-Tr2 50mcg; Drug: V3G CH848 Pr-NP1 100mcg
- Group 4: V3G CH848 Pr-NP1 with ACU-026-001-1 (Experimental): 3 doses of V3G CH848 Pr-NP1 (100 mcg) combined with ACU-026-001-1 (2.0 mg) at the month 0, 2, and 6 visits, followed by 1 dose of V3G CH848 mRNA-Tr2 (50 mcg) at the month 10 visit
  Interventions: Drug: V3G CH848 mRNA-Tr2 50mcg; Drug: ACU-026-001-1 2.0mg; Drug: V3G CH848 Pr-NP1 100mcg

INTERVENTIONS:
Drug: V3G CH848 Pr-NP1 60mcg — (60 mcg)
  Arms: Group 1: Low dose V3G CH848 Pr-NP1 with 3M-052-AF + Alum; Group 2: Low dose V3G CH848 Pr-NP1 with ACU-026-001-1
Drug: 3M-052-AF 5mcg — (5 mcg)
  Arms: Group 1: Low dose V3G CH848 Pr-NP1 with 3M-052-AF + Alum; Group 3: V3G CH848 Pr-NP1 with 3M-052-AF + Alum
Drug: Alum 500 mcg — (500 mcg)
  Arms: Group 1: Low dose V3G CH848 Pr-NP1 with 3M-052-AF + Alum; Group 3: V3G CH848 Pr-NP1 with 3M-052-AF + Alum
Drug: V3G CH848 mRNA-Tr2 50mcg — (50 mcg)
Drug: ACU-026-001-1 2.0mg — (2.0 mg)
  Arms: Group 2: Low dose V3G CH848 Pr-NP1 with ACU-026-001-1; Group 4: V3G CH848 Pr-NP1 with ACU-026-001-1
Drug: V3G CH848 Pr-NP1 100mcg — (100 mcg)
  Arms: Group 3: V3G CH848 Pr-NP1 with 3M-052-AF + Alum; Group 4: V3G CH848 Pr-NP1 with ACU-026-001-1

SUMMARY:
This first-in-human (FIH) phase 1 clinical trial will evaluate a prime-boost regimen of immunogens designed to induce HIV-1 Env V3-glycan-specific broadly neutralizing antibodies (V3G bNAbs). The priming immunogen (V3G CH848 Pr-NP1) consists of ferritin NPs expressing 8 copies of an Env trimer. This immunogen will be boosted with an mRNA LNP (V3G CH848 mRNA-Tr2), encoding a soluble Env trimer which does not utilize the ferritin NP design.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): Volunteer demonstrates an understanding of this study and completes a questionnaire prior to first vaccination with verbal demonstration of understanding of questionnaire items that were answered incorrectly.
* 18 to 55 years old, inclusive, on day of enrollment.
* Available for clinic follow-up through the last clinic visit, willing to undergo lymph node fine needle aspiration and leukapheresis, and willing to be contacted 12 months after the last study-product administration.
* Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 307 PSRT are required prior to enrollment into HVTN 307.
* In good general health according to the clinical judgment of the site investigator.
* Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
* Assessed by clinical staff as having a low likelihood of acquiring HIV per guidelines, agrees to discuss their potential for HIV acquisition, agrees to risk-reduction counseling, and agrees to avoid behaviors associated with a higher likelihood of acquiring HIV through the final study visit. Low likelihood may include persons stably taking pre-exposure prophylaxis (PrEP) as prescribed.
* Hemoglobin (Hgb):

  * ≥ 11.0 g/dL for volunteers AFAB
  * ≥ 13.0 g/dL for volunteers AMAB and for volunteers AFAB or intersex at birth who have been on masculinizing hormone therapy for more than 6 consecutive months
  * ≥ 12.0 g/dL for volunteers AMAB or intersex at birth who have been on feminizing hormone therapy for more than 6 consecutive months
  * For transgender or intersex volunteers who have been on hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth
* WBC count = 2,500 to 12,000/mm3 (WBC over 12,000/mm3 is not exclusionary if further evaluation shows general good health and if PSRT approval is granted).
* Platelets = 125,000 to 550,000/mm3.
* Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) based on the institutional normal range.
* Serum creatinine ≤ 1.1 x ULN based on the institutional normal range.
* A minimum limit of 8.5 mg/dL for corrected total serum calcium.
* Systolic blood pressure of 90 to <140 mmHg and diastolic blood pressure of 50 to <90 mmHg at screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mmHg systolic and 90 mmHg diastolic. A single measurement greater than or equal to 160 systolic mmHg or 100 mmHg diastolic during the current study evaluation is exclusionary.
* Negative HIV test results by one of the following options:

  * For US volunteers:
  * US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA)
  * Chemiluminescent microparticle immunoassay (CMIA)
  * Two negative results on HIV rapid tests (one of which must be FDA-approved CMIA)
* Negative for anti-Hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
* Negative for Hepatitis B surface antigen.
* For volunteers AFAB or intersex at birth and are of reproductive potential (hereafter referred to as "persons of pregnancy potential"):

  * Must agree to use effective means of birth control from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.
  * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.
* Volunteers of pregnancy potential must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

* Volunteer who is breastfeeding or pregnant.
* Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT approval.
* Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
* Previous or current recipient of an investigational HIV vaccine (previous placebo/ control recipients are not excluded).
* Receipt of non-HIV experimental vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) emergency use listing (EUL), or if outside the US, by the national Regulatory Authority (RA) authorizing this clinical trial.
* Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as glucocorticoid use, equal to or greater than prednisone 10 mg/day within 3 months prior to enrollment.
* Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
* Receipt of any of the following within 4 weeks prior to enrollment;

  * Live replicating vaccines
  * Any mRNA-based vaccine with FDA licensure, FDA emergency use authorization (EUA), or World Health Organization (WHO) emergency use listing
  * ACAM2000 vaccine > 28 days prior with a vaccination scab still present.
* Receipt of any vaccines that are not covered in #8 within 14 days prior to enrollment. Please note this includes replication incompetent vaccines such as the Jynneos vaccine for the prevention of mpox (formerly known as monkeypox) disease.
* Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
* Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
* History of serious reaction (eg, hypersensitivity, anaphylaxis) to any related vaccine or component of the study-vaccine regimen. Of note, the study proposed vaccine regimen includes components similar to components of the licensed COMIRNATY (Pfizer) and SPIKEVAX (Moderna) mRNA vaccines; severe reaction to these vaccines is therefore exclusionary.
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
* Idiopathic urticaria within the past year.
* Bleeding disorder diagnosed by a clinician which would make study procedures a contraindication.
* Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
* Asplenia or functional asplenia.
* Active duty and reserve US military personnel.
* Any other chronic or clinically significant condition that, in the clinical judgement of the investigator, would jeopardize the safety or rights of the study participant, including but not limited to: clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, persons with any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgement of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
* Asthma is excluded if the participant has ANY of the following:

  * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
  * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
  * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
  * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
  * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
* A participant with a history of a potential immune-mediated medical condition (PIMMC), either active or remote. Specific examples are listed in Appendix F (AESI Index). Not exclusionary: 1) Remote history of Bell's palsy (> 2 years ago) not associated with other neurologic symptoms and 2) mild psoriasis that does not require ongoing systemic treatment.
* History of allergy to local anesthetic (Novocaine, Lidocaine).
* Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.
* History of myocarditis and/or pericarditis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms for a minimum of 14 days following receipt of any study vaccine | 2 weeks following any injection
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Systemic reactogenicity signs and symptoms for a minimum of 14 days following receipt of any study vaccine. | 2 weeks following any injection
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Number of SAEs (Serious Adverse Events) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Number of MAAEs (medically attended adverse event) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Number of AESIs (Adverse events of special interest) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Number of AEs (adverse events) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Frequency of the V3G-specific precursor IgM+ and IgG+ B cells. | 2 weeks following injection
  Measured by flow cytometry analysis

SECONDARY OUTCOMES:
Response rate of serum IgG binding Abs | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by binding antibody multiplex assay (BAMA)
Magnitude of serum IgG binding Abs | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by binding antibody multiplex assay (BAMA)
Response rate of serum IgG binding Abs | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by BAMA
Magnitude of serum IgG binding Abs | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by BAMA
Response rate of serum Ab autologous neutralization of vaccine-matched tier 2 HIV-1 strains | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  measured by TZM-bl pseudovirus assay
Magnitude of serum Ab autologous neutralization of vaccine-matched tier 2 HIV-1 strains | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  measured by TZM-bl pseudovirus assay
Occurrence of CD4+ T-cell responses | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by intracellular cytokine staining in PMBCs
Magnitude of CD4+ T-cell responses | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by intracellular cytokine staining in PMBCs
Response rate of CD4+ T-cell responses | 2 weeks after the priming regimen and 2 weeks after the boost with V3G CH848 mRNA-Tr2
  Assessed by intracellular cytokine staining in PMBCs

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Alabama CRS [Site ID: 31788], Birmingham, Alabama
  - Emory University School of Medicine, The Ponce de Leon Center CRS [Site ID: 5802], Atlanta, Georgia
  - Brigham & Women's Hospital [Site ID: 30007], Boston, Massachusetts
  - BIDMC VCRS [Site ID: 32077], Boston, Massachusetts
  - Vanderbilt Vaccine (VV) CRS [Site ID: 30352], Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS [Site ID: 30331], Seattle, Washington

IPD SHARING:
Plan to Share IPD: No